CLINICAL TRIAL: NCT03360955
Title: Comparison of Extubation Time Between Total Intravenous Anesthesia Guided by Bispectral Index With Spinal Anesthesia With Minimal Opioid Dose for Cardiac Surgery
Brief Title: Comparison of Extubation Time Between Total Intravenous Anesthesia With Spinal Anesthesia for Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2017-3604-40
Record Dates: First submitted 2017-11-13; First posted 2017-12-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia
Keywords: Extubation; Cardiac Surgery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Intravenous Anesthesia: Patients with total intravenous anesthesia during the cardiac surgery
  Interventions: Procedure: Anesthesia
- Spinal Anesthesia: Patients with spinal anesthesia with minimal opioid dose.
  Interventions: Procedure: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia — Different anesthesia technique will be compared to find out which one offers better outcome to perform ultrafast track extubation

SUMMARY:
This study compares the extubation time between total intravenous anesthesia guided by Bispectral Index with spinal anesthesia with minimal opioid dose for cardiac surgery.

DETAILED DESCRIPTION:
This study compares the time needed to extubate of two anesthesic techniques, 1) Total Intravenous Anesthesia guided by Bispectral Index (BIS), 2) Spinal Anesthesia with minimal opioid dose for cardiac surgery.

Identify the best anesthesia technique to do ultrafast track extubation can minimize the risk of infection associated.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for cardiac surgery Physical Status Classification System of the American Society of Anesthesiologists (ASA) II-III

Exclusion Criteria:

Physical Status Classification System of the American Society of Anesthesiologists (ASA) IV-V Emergency cardiac surgery Spinal defect

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Extubation time | Up to 1 hour after anesthesia emergence
  The time from anesthesia emergence to extubation will be measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gabriela Gallardo, PhD, Principal Investigator — IMSS
Locations (1):
- Hospital de cardiología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided